CLINICAL TRIAL: NCT04340310
Title: Usefulness of Home Respiratory Polygraphy in the Diagnosis and Therapeutic Decision of Childhood Sleep Apnea-Hypopnea Syndrome
Brief Title: Home Respiratory Polygraphy in Childhood Sleep Apnea-Hypopnea Syndrome (CHILDSLEEP).
Acronym: CHILDSLEEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Principal Investigator, Eusebi Chiner, Head of Pneumology, Hospital Universitario San Juan de Alicante
Other Study IDs: CEIC (HUSJ-20-003)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Sleep Apnea; Home Respiratory Polygraphy Sleep Study; Childhood Sleep Apnea; Polysomnography; Therapeutic Decision
Keywords: Childhood sleep apnea; Sleep apnea syndrome; Obstructive apnea syndrome; Obstructive apnea sleep
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home respiratory poligraphy: Group A: Children between 4 and 14 years-old with initial OSA suspicion there will be allocated to Home Respiratory Polygraphy (HRP)
  Interventions: Diagnostic Test: Home respiratory polygraphy
- Polysomnography: Group B: Children between 4 and 14 years-old with initial OSA suspicion and concommitant diseases and false negative suspicion from HRP there will allocated to Hospital Nocturnal Polysomnography
  Interventions: Diagnostic Test: Home respiratory polygraphy

INTERVENTIONS:
Diagnostic Test: Home respiratory polygraphy — Home respiratory polygraphy or Polysomnography to stablish a therapeutic decission
  Other Names: Polysomnography

SUMMARY:
The aims of the study is to assess the diagnostic utility of home respiratory polygraphy (HRP) complemented with polysomnography (PSG) in childhood Obstructive Sleep Apnea-Hypopnea Syndrome (OSAS), as well as its usefulness in the therapeutic decisions.

Methods: Children referred with suspected OSAS will be evaluated during one year performing home respiratory polygraphy in all cases. PSG will be chosen in patients with concomitant pathology or according to medical criteria, or complemented with HRP in doubtful cases. Clinical and anthropometric data, severity, technical quality and treatment will be obtained. Patients will be divided in two groups (HRP vs PSG) and compared, and the accuracy from HRP to establish a therapeutic decision it wil calculated. The investigator's hypothesis is that PSG should be recommended only for complex or doubtful cases.

ELIGIBILITY:
Inclusion Criteria:

* Sleep apnea suspicion

Exclusion Criteria:

* Other sleep conditions
* Non valid home respiratory polygraphy and non valid polysomnography in the same patient
* Non informated consent

Ages: 4 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Children submited to Pneumology Service with sleep apnea suspicion
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-04-06 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic utility of home respiratory polygraphy (HRP) complemented with polysomnography (PSG) in childhood Obstructive Sleep Apnea-Hypopnea Syndrome (OSAS), as well as its usefulness in the therapeutic decisions. | two years
  False negative and true positive diagnosis by home respiratory polygraphy

SECONDARY OUTCOMES:
To assess the prevalence of childhood sleep apnea in Pneumology hospital consultations | two years
  Number of chlidhood sleep consultations related to adult consultations

CONTACTS AND LOCATIONS:
Overall Officials: Eusebi Chiner Vives, Principal Investigator — Hospital Universitario San Juan de Alicante
Locations (1):
- Eusebio Chiner Vives, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
Scientific publication, Sleep spanish network
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years